CLINICAL TRIAL: NCT00859066
Title: Evaluation of Radiology Resident Anxiety When Beginning ER Call
Brief Title: Evaluation of Radiology Resident Anxiety When Beginning Emergency Room (ER) Call
Status: Terminated | Type: Observational
Why Stopped: Original Principal Investigator (Andrew Trout M.D.) left the University.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Richard Cohan M.D., Principal Investigator, University of Michigan
Other Study IDs: HUM00026874
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Anxiety; Stress
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control Group: First year University of Michigan Radiology residents will take call as scheduled without a "buddy call" experience.
  (Enrollment completed for the control group)
- Experimental Group: 2009 class of first year Radiology residents who will be assigned two 5 hour shifts working side by side with a more senior resident (who has experience taking call).

SUMMARY:
The purpose of this study is to quantify levels of resident anxiety under the current system (take call alone) and compare results to a modified system.

DETAILED DESCRIPTION:
The study purpose is to quantify resident perceptions and feelings under the current 1700 call system (take call alone) and compare those with resident perceptions and feelings under a modified system where two partial shifts are taken with an experienced resident ("buddy call") prior to taking call alone.

ELIGIBILITY:
Inclusion Criteria:

* first year radiology residents

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: First year radiology residents
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improve resident well-being by decreasing anxiety surrounding beginning ER call as a first year radiology resident. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cohan, M.D., Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States